CLINICAL TRIAL: NCT00197730
Title: Trial of Vitamins Among Children of HIV-infected Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Wafaie Fawzi, Harvard School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HD43688
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: HIV Infections; Pregnancy Complications
Keywords: Birth Outcomes; Nutrition; HIV; AIDS; Vitamins; Multivitamins; Maternal and child health outcomes; Tanzania; Africa
MeSH Terms: conditions — HIV Infections; Pregnancy Complications; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multivitamins (Experimental): Vitamin E, Vitamin C, and Vitamin B complex
  Interventions: Drug: Multivitamins - vitamins B complex, C and E
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Multivitamins - vitamins B complex, C and E — Age-appropriate dosages of vitamin C, vitamin E, thiamine, riboflavin, niacin, vitamin B6, folate, and vitamin B12 administered orally to children aged 6 weeks to 6 months, and two capsules per day for children aged older than 6 months for at least 12 months
  Arms: Multivitamins
Drug: Placebo — Placebo capsules administered orally once day orally to children aged 6 weeks to 6 months, and twice per day for children aged older than 6 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effects of multivitamin (B, C, E) supplementation on reducing the risk of morbidity and mortality outcomes among children born to HIV positive mothers, compared to placebo supplementation.

DETAILED DESCRIPTION:
An increasing body of evidence supports the efficacy of single and, more recently, multiple micronutrient supplementation in reducing morbidity and mortality in susceptible populations. For example, we recently completed a multiple micronutrient supplementation trial in HIV-positive Tanzanian women that showed a significant reduction in pre-term birth, fetal loss, and low birthweight. In children, we and others have also demonstrated the beneficial effects of vitamin A supplementation in reducing diarrheal disease and mortality. Our next priority is to evaluate the efficacy of multiple micronutrient supplementation in susceptible children. Children born to HIV-infected women are at risk of multiple micronutrient deficiencies due to poor dietary intake, malabsorption, and increased metabolic needs. In addition, these children, if HIV-infected themselves, are at significantly higher risk of death due to infectious illnesses compared to their non-infected peers. In this study, we propose to study the efficacy of micronutrient supplementation in reducing the risk of morbidity and mortality outcomes among children born to HIV positive mothers, compared to placebo supplementation.

ELIGIBILITY:
Inclusion Criteria: Singleton, live born infants born to HIV-infected women Exclusion Criteria: Infants with multiple congenital abnormalities

Ages: 6 Weeks to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2387 (Actual)
Dates: Start 2004-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
All-cause mortality and diarrheal morbidity | age 6 weeks to age 24 months

SECONDARY OUTCOMES:
Child growth faltering, lower respiratory infections, HIV breastfeeding transmission, and maternal HIV disease progression in relation to breastfeeding | age 6 weeks to 24 months post partum

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, MD, DrPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

REFERENCES:
- [Derived] Rees CA, Kisenge R, Manji KP, Liu E, Fawzi WW, Duggan CP. Identifying Infants and Young Children at Risk of Unplanned Hospital Admissions and Clinic Visits in Dar es Salaam, Tanzania. Pediatr Infect Dis J. 2020 Dec;39(12):e428-e434. doi: 10.1097/INF.0000000000002875. PMID 32842043
- [Derived] Blakstad MM, Smith ER, Etheredge A, Locks LM, McDonald CM, Kupka R, Kisenge R, Aboud S, Bellinger D, Sudfeld CR, Fawzi WW, Manji K, Duggan CP. Nutritional, Socioeconomic, and Delivery Characteristics Are Associated with Neurodevelopment in Tanzanian Children. J Pediatr. 2019 Apr;207:71-79.e8. doi: 10.1016/j.jpeds.2018.10.066. Epub 2018 Dec 14. PMID 30559023
- [Derived] Locks LM, Mwiru RS, Mtisi E, Manji KP, McDonald CM, Liu E, Kupka R, Kisenge R, Aboud S, Gosselin K, Gillman M, Gewirtz AT, Fawzi WW, Duggan CP. Infant Nutritional Status and Markers of Environmental Enteric Dysfunction are Associated with Midchildhood Anthropometry and Blood Pressure in Tanzania. J Pediatr. 2017 Aug;187:225-233.e1. doi: 10.1016/j.jpeds.2017.04.005. Epub 2017 May 9. PMID 28499715
- [Derived] Locks LM, Manji KP, Kupka R, Liu E, Kisenge R, McDonald CM, Aboud S, Wang M, Fawzi WW, Duggan CP. High Burden of Morbidity and Mortality but Not Growth Failure in Infants Exposed to but Uninfected with Human Immunodeficiency Virus in Tanzania. J Pediatr. 2017 Jan;180:191-199.e2. doi: 10.1016/j.jpeds.2016.09.040. Epub 2016 Nov 7. PMID 27829511
- [Derived] Sztam KA, Liu E, Manji KP, Kupka R, Kisenge R, Aboud S, Fawzi WW, Bosch RJ, Duggan CP. Maternal Antiretroviral Therapy Is Associated with Lower Risk of Diarrhea in Early Childhood. J Pediatr. 2016 Aug;175:54-60. doi: 10.1016/j.jpeds.2016.04.088. Epub 2016 May 28. PMID 27245295
- [Derived] Manji KP, Duggan C, Liu E, Bosch R, Kisenge R, Aboud S, Kupka R, Fawzi WW. Exclusive Breast-feeding Protects against Mother-to-Child Transmission of HIV-1 through 12 Months of Age in Tanzania. J Trop Pediatr. 2016 Aug;62(4):301-7. doi: 10.1093/tropej/fmw012. Epub 2016 Mar 15. PMID 26999011
- [Derived] Sudfeld CR, Duggan C, Aboud S, Kupka R, Manji KP, Kisenge R, Fawzi WW. Vitamin D status is associated with mortality, morbidity, and growth failure among a prospective cohort of HIV-infected and HIV-exposed Tanzanian infants. J Nutr. 2015 Jan;145(1):121-7. doi: 10.3945/jn.114.201566. Epub 2014 Nov 12. PMID 25527666
- [Derived] Sudfeld CR, Duggan C, Histed A, Manji KP, Meydani SN, Aboud S, Wang M, Giovannucci EL, Fawzi WW. Effect of multivitamin supplementation on measles vaccine response among HIV-exposed uninfected Tanzanian infants. Clin Vaccine Immunol. 2013 Aug;20(8):1123-32. doi: 10.1128/CVI.00183-13. Epub 2013 May 29. PMID 23720367
- [Derived] Kupka R, Manji KP, Bosch RJ, Aboud S, Kisenge R, Okuma J, Fawzi WW, Duggan C. Multivitamin supplements have no effect on growth of Tanzanian children born to HIV-infected mothers. J Nutr. 2013 May;143(5):722-7. doi: 10.3945/jn.112.170498. Epub 2013 Mar 20. PMID 23514773
- [Derived] Duggan C, Manji KP, Kupka R, Bosch RJ, Aboud S, Kisenge R, Okuma J, Fawzi WW. Multiple micronutrient supplementation in Tanzanian infants born to HIV-infected mothers: a randomized, double-blind, placebo-controlled clinical trial. Am J Clin Nutr. 2012 Dec;96(6):1437-46. doi: 10.3945/ajcn.112.044263. Epub 2012 Nov 7. PMID 23134887
- [Derived] McDonald CM, Kupka R, Manji KP, Okuma J, Bosch RJ, Aboud S, Kisenge R, Spiegelman D, Fawzi WW, Duggan CP. Predictors of stunting, wasting and underweight among Tanzanian children born to HIV-infected women. Eur J Clin Nutr. 2012 Nov;66(11):1265-76. doi: 10.1038/ejcn.2012.136. Epub 2012 Oct 3. PMID 23031850